CLINICAL TRIAL: NCT06642623
Title: A Prospective, Open, Registry-based Randomized, Controlled, Investigator Initiated Trial of Enavogliflozin(ENVlo) to EvaLuate Cardio-renal Outcome in Type 2 Diabetes Mellitus Patients (ENVELOP Study)
Brief Title: A Prospective Trial of Enavogliflozin to Evaluate Cardio-renal Outcome in Type 2 Diabetes Mellitus Patients
Acronym: ENVELOP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-1334
Record Dates: First submitted 2024-10-13; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases; Kidney Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Kidney Diseases | interventions — Enavogliflozin; dapagliflozin; empagliflozin

STUDY DESIGN:
Intervention Model Description: his study was designed as a pragmatic clinical trial(pracmatic RCT), which demonstrates the real-world effectiveness of the intervention in broad patient groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enavogliflozin Group (Experimental): Subjects will take Enavogliflozin according to the investigator's judgment.
  Interventions: Drug: Enavogliflozin
- Dapagliflozin, Empagliflozin Group (Active Comparator): Subjects will take Dapagliflozin or Empagliflozin according to the investigator's judgment.
  Interventions: Drug: Dapagliflozin or Empagliflozin

INTERVENTIONS:
Drug: Enavogliflozin — The dosage and administration method are determined according to the investigator's judgment, considering the drug's approval requirements and the medical condition of the study participants.
  Arms: Enavogliflozin Group
Drug: Dapagliflozin or Empagliflozin — The dosage and administration method are determined according to the investigator's judgment, considering the drug's approval requirements and the medical condition of the study participants.
  Arms: Dapagliflozin, Empagliflozin Group

SUMMARY:
The novel sodium-glucose cotransporter-2 (SGLT2) inhibitor, enavogliflozin, effectively reduces glycated hemoglobin (HbA1c) levels and body weight without increasing the risk of serious adverse events. However, its long-term clinical benefits concerning cardiovascular and renal outcomes have yet to be thoroughly studied. This study is an investigator-initiated, multicenter, randomized, pragmatic, open-label, active-controlled, non-inferiority trial. Eligible participants are adults aged 19 or older with type 2 diabetes who have a history of, or are at risk for, cardiovascular disease. A total of 2,862 participants will be randomly assigned to receive either enavogliflozin or other SGLT2 inhibitors with proven cardiorenal benefits, such as dapagliflozin or empagliflozin. The primary endpoint is the time to the first occurrence of a composite of major adverse cardiovascular and renal events. This trial aims to determine whether enavogliflozin is non-inferior to dapagliflozin or empagliflozin in terms of cardiorenal outcomes in patients with type 2 diabetes and cardiovascular risk factors. It will also clarify role of enavogliflozin in preventing vascular complications in this patient population.

DETAILED DESCRIPTION:
The ENVELOP study aims to assess cardiorenal outcomes following enavogliflozin administration compared with dapagliflozin or empagliflozin in Korean patients with type 2 diabetes, representing the first large-scale SGLT2 inhibitor outcome study targeting this population.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults aged 19 years and older at screening
2. Subjects diagnosed with T2D at screening
3. Subjects on treatment with or requiring treatment with enavogliflozin, dapagliflozin, or empagliflozin within the scope of label and reimbursement criteria

Exclusion Criteria:

1. Subjects with different types of diabetes mellitus other than T2D
2. Subjects with moderate to severe hepatic impairment
3. Subjects with contraindications to SGLT-2 inhibitors, i.e., kidney function disorders with estimated glomerular filtration (eGFR) <60 mL/min/1.73 m2, end stage renal disease (ESRD), or on dialysis
4. Subjects with major comorbidities
5. Subjects with a history of hypersensitivity to enavogliflozin, dapagliflozin, or empagliflozin and any of its components
6. Pregnant or breastfeeding women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2862 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Time from randomization to first onset of cardiorenal composite outcome event | 6 months, 12 months, 24 months, 36 months and 48 month
  Major adverse cardiovascular events include nonfatal myocardial infarction (MI), nonfatal stroke, and hospitalization for unstable angina, hospitalization for heart failure, coronary or peripheral revascularization, and death from any cause. Renal events include a sustained decline in estimated glomerular filtration rate (GFR) calculated by means of the Chronic Kidney Disease Epidemiology Collaboration equation of ≥40% from baseline to <60 mL/min/1.73m2, onset of end-stage kidney disease (dialysis for ≥28 days, kidney transplantation, or an estimated GFR of <15 mL/min/1.73m2), development of macroalbuminuria, and death from renal causes.

SECONDARY OUTCOMES:
Time from randomization to the first onset of 3-point MACE and proportion of the patients | 6 months, 12 months, 24 months, 36 months and 48 months
  Time to first event of a composite of key major adverse cardiovascular events (non-fatal MI, non-fatal stroke, and death from cardiovascular causes)
death from any cause | 6 months, 12 months, 24 months, 36 months and 48 months
  Time to death from any cause
death from cardiovascular causes | 6 months, 12 months, 24 months, 36 months and 48 months
  Time to death from cardiovascular cause
hospitalization due to unstable angina | 6 months, 12 months, 24 months, 36 months and 48 months
  Time to first event of hospitalization due to unstable angina
hospitalization due to heart failure | 6 months, 12 months, 24 months, 36 months and 48 months
  Time to first event of hospitalization due to heart failure
coronary or peripheral revascularization | 6 months, 12 months, 24 months, 36 months and 48 months
  Time to first event of coronary or peripheral revascularization
major renal events | 6 months, 12 months, 24 months, 36 months and 48 months
  Time to first event of a composite of major kidney events
progression of macroalbuminuria | 6 months, 12 months, 24 months, 36 months and 48 months
  Time to development of macroalbuminuria

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine, 50-1 Yonsei-ro, Seodaemun-gu, Seoul 03722, Republic of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No